CLINICAL TRIAL: NCT02634476
Title: Can Cognitive-bias Modification Training During Inpatient Alcohol Detoxification Reduce Relapse Rates Post-discharge?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turning Point (Other)
Collaborators: Monash University (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E33-1314
Record Dates: First submitted 2015-10-16; First posted 2015-12-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Dependence
Keywords: Alcohol; Substance use disorder; cognitive bias; behavioral intervention; computerised training
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive bias modification training (Experimental): Participants complete four sessions of the alcohol approach/avoidance task.
  Interventions: Behavioral: Alcohol approach/avoidance task
- sham training (Sham Comparator): Participants complete four sessions of the sham approach/avoidance task.
  Interventions: Behavioral: Sham approach/avoidance task

INTERVENTIONS:
Behavioral: Alcohol approach/avoidance task — The approach-bias modification is a computerised alcohol approach/avoidance task (alcohol-AAT) in which participants are instructed to respond with an approach movement (pulling a joystick) to pictures in landscape orientation and an avoidance movement (pushing a joystick) to pictures in portrait orientation. The size of the image is increased and decreased by pulling and pushing the joystick respectively, generating a sensation of approach or avoidance. Pictures include images of 20 alcoholic and 20 non-alcoholic drinks presented in a fixed orientation such that participants are in effect instructed to respond to pictures of alcohol by making an avoidance movement (pushing the joystick) and to pictures of non-alcoholic soft drinks by making an approach movement (pulling the joystick).
  Other Names: Alcohol-AAT; Alcohol cognitive bias modification training
  Arms: cognitive bias modification training
Behavioral: Sham approach/avoidance task — The computerised training for the sham condition is the same as for the experimental condition, except that in the sham approach/avoidance task, both landscape and portrait pictures all contain neutral (non-alcohol related).
  Other Names: Sham-AAT; Sham cognitive bias modification training
  Arms: sham training

SUMMARY:
It is well-established that many substance misusers experience impairment in cognition (thinking skills), particularly those needed to regulate and monitor behaviour and ensure that goals are achieved. According to the dual-process model, addiction arises from an imbalance in 'bottom-up' processing i.e., overactive automatic (impulsive) processes that drive behaviours and impaired 'top-down' controlling processes that stop behaviours associated with negative consequences. As a result, the individual becomes more sensitive to cues in their environment (e.g., alcohol images) that trigger the addictive behaviour. Cognitive-bias modification (CBM) is a novel, computer-based training paradigm that trains the brain to pay less attention to negative/harmful cues and more attention to positive or neutral cues. This approach minimizes the overactive 'bottom-up' processes and improves the 'top-down' control processes of unhealthy behaviors which enables the addicted individual to make better decisions. Recently, CBM has been used with addicted population to alter the tendency to approach alcohol, with one German study showing that a 4-session training programme was associated higher rates of abstinence at one-year (Wiers et al., 2011). The current study examines whether a novel computer based training programme alters cognitive biases (the tendency to approach alcohol related stimuli) in alcohol-dependent inpatients, and examine whether this enables them to be better at decision-making more generally, and its impact on craving and post-discharge abstinence rates. The study will also explore whether individual differences in impulsivity and sensitivity to reward and punishment determine response to the training programme. This will be achieved using a parallel-groups randomized superiority trial design involving approximately 80 patients attending inpatient withdrawal programmes in Victoria. The findings are likely to have implications for the design and delivery of psychosocial interventions delivered during early recovery from alcohol-dependence to optimise treatment effectiveness.

DETAILED DESCRIPTION:
Detailed Description:

According to the dual-process model of addiction (Gullo, Loxton, & Dawe, 2014), addictive behaviour is the result of an imbalance between a strong, impulsive processing system and a relatively weak, reflective processing system. Due to this imbalance, impulsive preferences are rewarded, reflected in an increased sensitivity to the stimuli of addiction (i.e., attentional bias) and an automatic tendency to engage with the stimuli of addiction (i.e., approach bias; Wiers et al., 2007). Clinical trials of CBM have begun to emerge for individuals with alcohol use disorders (Fadardi & Cox, 2009). Wiers et al. (2009) developed the alcohol approach/avoidance task (alcohol-AAT), where participants respond with an approach behaviour (pulling a joystick) or an avoidance behaviour (pushing a joystick) to pictures of addiction-related and neutral stimuli. Following four sessions of this training task patients displayed better treatment outcomes one-year later (Wiers et al., 2011). A study by Eberl et al. (2013) found that 12 sessions of approach-bias modification training was associated with higher rates of abstinence at one-year relative to controls.

Underlying the relationship between cognitive biases and addiction, within the dual-process model paradigm, are impulse-control processes. However, the relationship between impulsivity and cognitive biases remains unclear. Indeed, individuals with weak inhibition skills tend to have a bias toward automatic information processing (Gladwin et al., 2011) and impulsivity is thought to play a role in the degree to which cognitive biases influence outcomes (Peeters et al., 2012). The development of this understanding will benefit assessment of CBM treatments for addiction patients.

Rationale:

Despite intensive psychosocial interventions, most alcohol-dependent patients relapse within weeks if not days of leaving inpatient detoxification. The study therefore examines whether an alcohol approach-bias modification training programme during detox can reduce craving and relapse in alcohol-dependent inpatients. By dampening the automatic tendency to approach alcohol-related stimuli, individuals are allowing time to make more informed behaviour choices (i.e., improving their decision-making ability). Its impact will be examined through abstinence rates at 2-weeks and 3-months relative to those receiving sham training. The findings are likely to have implications for the design and delivery of psychosocial interventions delivered during early recovery from alcohol-dependence, aiming to optimise treatment effectiveness.

Aims:

1. To determine if 4-sessions of CBM, using an alcohol approach-bias modification training program, delivered during inpatient withdrawal, reduces craving and relapse rates and other drinking-related outcomes at 2-weeks and 3-months post-discharge.
2. To determine if CBM, using alcohol approach-bias modification training, improves decision-making after four training sessions.
3. To determine if CBM effects (i.e., using alcohol approach-bias modification training) are moderated by impulsivity.

Hypotheses:

1. CBM (using alcohol approach-bias modification training) will lead to significantly higher rates of abstinence at 2-weeks and 3-months and larger reductions in days to relapse, percentage of heavy drinking days and craving score, relative to sham training.
2. CBM (using alcohol approach-bias modification training) will be associated with significantly greater improvement in decision-making (Iowa Gambling Task performance) after the fourth training session compared to sham training.
3. Patients with greater impulsivity will show significantly greater responses to CBM (using alcohol approach-bias modification training).

Methodology:

The study will be a parallel-groups randomized superiority trial comparing CBM (using alcohol approach-bias modification training) versus sham training (i.e., control condition) in alcohol-dependent participants following residential detoxification treatment. The primary outcome variables will be self-reported alcohol use (relapse versus abstinence) 2-weeks and 3-months post discharge and secondary outcomes will include: days to relapse, percentage of heavy drinking days, alcohol craving and Iowa Gambling Task performance (i.e., decision-making) immediately post-intervention.

Assignment:

Randomisation will be carried out according to the ICH Guideline by an independent statistician not involved in the day-to-day conduct of the trial. Following baseline assessments, participants will be assigned randomly to the treatment condition using a 1:1 ratio and randomly permuted blocks.

Participants:

The target sample is defined as alcohol-dependent patients seeking treatment at the detoxification inpatient unit in Wellington House, Box Hill, Victoria.

Setting:

Wellington House, an inpatient detoxification service; part of Turning Point, a state-wide Alcohol and other Drug (AOD) service that incorporates Eastern region based services.

Measures:

Standard demographic questionnaire including: age, gender, history of alcohol use, previous alcohol treatment, employment, income source, housing arrangements, family situation, mental health. Current medication regimen, including psychotropic medications. All benzodiazepines will be converted to standard dose of diazepam.

Baseline drug use and clinical measures:

Alcohol/Drug use: Timeline Followback Interview (TLFB; Sobell & Sobell, 1992): as a measure of frequency of alcohol/drug use in the past 4 weeks.

Baseline alcohol dependence: Severity of Alcohol Dependence Questionnaire (SADQ; Stockwell et al, 1983).

General cognitive functioning: Montreal Cognitive Assessment (MoCA): a brief cognitive screening tool of general cognitive functioning (Nasreddine et al, 2005).

Appetitive motivational behaviour/ impulsivity: The Sensitivity to Reward (SR) part of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ; Torrubia et. al., 2001); specifically measures appetitive motivational behaviour or impulsivity.

Impulsiveness, venturesomeness, empathy: The I7 Impulsiveness questionnaire (Eysenck, Pearson, Easting & Allsopp, 1985) is a 54-item measure consisting of three scales: impulsiveness, venturesomeness, and empathy.

Craving: Assessed using 100mm visual analogue scales (VAS). The VAS provides an index of urge to drink using two dimensions (positive and negative urge; Dawe & Gray, 1995).

Craving: The Alcohol Craving-Short-Form-Revised (ACQ-SF-R: Singleton, 2000) is a 12-item measure of craving for alcohol among alcohol users in the current context (right now).

Depression and anxiety: Seven depression and seven anxiety items of the shortened Depression Anxiety and Stress Scale (DASS; Lovibond & Lovibond, 1995).

Decision-making: A computerised version of the Iowa Gambling Task (IGT; Bechara et al., 2000): measures decision-making under conditions of uncertainty and risk of punishment.

Procedures:

Recruitment and consent: Participants will be approached by a researcher no earlier than day three of admission. All Participants will be provided with a Plain Language statement explaining the purpose of the study and what will be required of participants. The study will also be explained verbally by the researchers. If the participant chooses to become part of the study a written consent form (i.e., Patient Information and Consent Form) will be completed. The researcher will also seek consent to contact others and document relevant telephone/contact details so that self-reported outcome can be assessed 2-weeks and 3-months post-discharge.

Baseline, intervention and post-intervention outcome assessment: Following the consent taking, the baseline assessment will be completed as described in the measures section. Participants will then be randomised to one of two conditions, cognitive bias training or sham training. On the morning of days 3/4 to days 6/7 (i.e., four consecutive days) of admission, participants will undergo the ABM (intervention). Each training session is expected to last approximately 15 minutes. Participants will be given the opportunity to take an optional break during the intervention. After the final (i.e., fourth) training session, participants will complete the post training assessment (decision-making task and craving measures).

Two-weeks and 3 months post discharge the researcher will telephone the participant to use the timeline follow-back instrument to document alcohol consumption since discharge and ask questions about engagement in treatment since discharge.

Statistical Analyses:

The primary hypothesis uses a binary outcome variable (abstinent versus relapse at 2-weeks) following completion of the protocol (four sessions) and will be examined using chi-square analyses. Secondary outcomes which are continuous variables (i.e., days to relapse, percentage of heavy drinking days, mean number of standard drinks, craving scores, IGT score etc.) will be examined using mixed effects repeated measures models (MMRM) including type of intervention (cognitive bias modification training versus sham training) as the independent variable and craving, decision-making, days to relapse and other alcohol consumption outcomes as dependent variables. The third hypothesis will be tested with a multiple regression model including sensitivity to reward and impulsivity scores at baseline, as predictors of outcome (abstinence, days to relapse etc..). Power calculations based on a hypothesized medium effect size indicate that a sample size of 72 participants (36 in each group) is required to test the study hypotheses with 80% power.

ELIGIBILITY:
Inclusion Criteria:

* At least weekly use of alcohol in the past month.
* Meet Diagnostic and Statistical Manual (DSM) criteria for alcohol use disorder
* Currently in treatment for alcohol withdrawal
* Able to understand English

Exclusion Criteria:

* Meet Diagnostic and Statistical Manual (DSM) criteria for a psychotic illness
* History of neurological illness
* History of brain injury involving loss of consciousness for >30 minutes
* Intellectual disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Alcohol abstinence | 2-week follow-up
  We will assess whether the participant has consumed alcohol at any time between exiting the detoxification facility and completing the 2-week follow-up questionnaires.

SECONDARY OUTCOMES:
Days until relapse | 2-week follow-up
  In those who drink before the 2-week follow-up, we will assess the number of days between discharge from detoxification and their first drink of alcohol.
Number of heavy drinking days | 2-week follow-up
  We will assess the number of days, in the 14 days prior to the 2-week follow-up, on which the participant consumed at least 5 standard drinks of alcohol.
Alcohol craving | Immediately after the 4th training session (days 6 or 7 following admission)
  We will assess craving for alcohol following the final session with both a visual analogue scale and the Alcohol Craving Questionnaire (Short Form - Revised).
Alcohol craving | 2-week follow-up
  We will assess craving for alcohol following the final session with the Alcohol Craving Questionnaire (Short Form - Revised).
Abstinence at 3-months | 3-month follow-up
  We will assess whether the participant has consumed alcohol at any time during the 30 days prior to the 3-month follow-up.
Decision-making | Immediately after the 4th training session (days 6 or 7 following admission)
  The Iowa Gambling Task will be administered following the final training session.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Manning, PhD, Principal Investigator — Senior Research Fellow
Locations (1):
- Wellington House, Box Hill, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338
- [Background] Eberl C, Wiers RW, Pawelczack S, Rinck M, Becker ES, Lindenmeyer J. Implementation of approach bias re-training in alcoholism-how many sessions are needed? Alcohol Clin Exp Res. 2014 Feb;38(2):587-94. doi: 10.1111/acer.12281. Epub 2013 Oct 24. PMID 24164417
- [Background] Gladwin TE, Figner B, Crone EA, Wiers RW. Addiction, adolescence, and the integration of control and motivation. Dev Cogn Neurosci. 2011 Oct;1(4):364-76. doi: 10.1016/j.dcn.2011.06.008. Epub 2011 Jul 2. PMID 22436562
- [Background] Bechara A, Tranel D, Damasio H. Characterization of the decision-making deficit of patients with ventromedial prefrontal cortex lesions. Brain. 2000 Nov;123 ( Pt 11):2189-202. doi: 10.1093/brain/123.11.2189. PMID 11050020
- [Background] Dawe S, Gray JA. Craving and drug reward: a comparison of methadone and clonidine in detoxifying opiate addicts. Drug Alcohol Depend. 1995 Oct;39(3):207-12. doi: 10.1016/0376-8716(95)01159-8. PMID 8556969
- [Background] Fadardi JS, Cox WM. Reversing the sequence: reducing alcohol consumption by overcoming alcohol attentional bias. Drug Alcohol Depend. 2009 May 1;101(3):137-45. doi: 10.1016/j.drugalcdep.2008.11.015. Epub 2009 Feb 3. PMID 19193499
- [Background] Gullo MJ, Loxton NJ, Dawe S. Impulsivity: four ways five factors are not basic to addiction. Addict Behav. 2014 Nov;39(11):1547-1556. doi: 10.1016/j.addbeh.2014.01.002. Epub 2014 Jan 16. PMID 24576666
- [Background] Peeters M, Wiers RW, Monshouwer K, van de Schoot R, Janssen T, Vollebergh WA. Automatic processes in at-risk adolescents: the role of alcohol-approach tendencies and response inhibition in drinking behavior. Addiction. 2012 Nov;107(11):1939-46. doi: 10.1111/j.1360-0443.2012.03948.x. Epub 2012 Aug 28. PMID 22632107
- [Background] Wiers RW, Rinck M, Dictus M, van den Wildenberg E. Relatively strong automatic appetitive action-tendencies in male carriers of the OPRM1 G-allele. Genes Brain Behav. 2009 Feb;8(1):101-6. doi: 10.1111/j.1601-183X.2008.00454.x. Epub 2008 Nov 11. PMID 19016889
- [Background] Eberl C, Wiers RW, Pawelczack S, Rinck M, Becker ES, Lindenmeyer J. Approach bias modification in alcohol dependence: do clinical effects replicate and for whom does it work best? Dev Cogn Neurosci. 2013 Apr;4:38-51. doi: 10.1016/j.dcn.2012.11.002. Epub 2012 Nov 14. PMID 23218805
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Wiers RW, Bartholow BD, van den Wildenberg E, Thush C, Engels RC, Sher KJ, Grenard J, Ames SL, Stacy AW. Automatic and controlled processes and the development of addictive behaviors in adolescents: a review and a model. Pharmacol Biochem Behav. 2007 Feb;86(2):263-83. doi: 10.1016/j.pbb.2006.09.021. Epub 2006 Nov 20. PMID 17116324
- [Derived] Manning V, Staiger PK, Hall K, Garfield JB, Flaks G, Leung D, Hughes LK, Lum JA, Lubman DI, Verdejo-Garcia A. Cognitive Bias Modification Training During Inpatient Alcohol Detoxification Reduces Early Relapse: A Randomized Controlled Trial. Alcohol Clin Exp Res. 2016 Sep;40(9):2011-9. doi: 10.1111/acer.13163. Epub 2016 Aug 4. PMID 27488392
- See also: Sobell, LC.; Sobell, MB. Timeline follow-back: A technique for assessing self-reported alcohol consumption. In: Raye, Z.; Litten, JPA., editors. Measuring alcohol consumption: Psychosocial and biochemical methods. Totowa, NJ: Humana Press, Inc; 1992 — http://link.springer.com/chapter/10.1007/978-1-4612-0357-5_3#page-1
- See also: Singleton, E.G., Tiffany, S.T. & Henningfield, J.E. (2000). Alcohol Craving — http://adai.washington.edu/instruments/pdf/Alcohol_Craving_Questionnaire_Short_Form_Revised_20.pdf
- See also: Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety Stress Scales. (2nd. Ed.) Sydney: Psychology Foundation. — http://www2.psy.unsw.edu.au/dass/